CLINICAL TRIAL: NCT01550133
Title: Effects of Nutritive and Non-Nutritive Food Form and Learning on Cephalic Phase Responses
Brief Title: Effects of Food Form on Cephalic Phase Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R01DK079913-4; R01DK079913 (NIH); 1201011780 (Other: Purdue University)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Obese; Overweight
Keywords: Peptides; Hormones; Appetite; Humans; Obese; Beverage; Solid food; cephalic phase
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Not Learned: Non-nutritive bev to Nutritive bev (Experimental): 15 participants will be randomly assigned to eat 250 grams of non-nutritive solid consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a nutritive solid and act as a control for the learned effects.
  Interventions: Behavioral: Learned: Non-nutritive beverage to Non-nutritive beverage
- Not Learned: Nutritive solid to Non-Nutritive solid (Experimental): 15 participants will be randomly assigned to eat 250 grams of nutritive solid consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a non-nutritive solid and act as a control for the learned effects.
  Interventions: Behavioral: Learned: Nutritive solid to Nutritive solid
- Not Learned: Nutritive beverage to Non-Nutritive beverage (Experimental): 15 participants will be randomly assigned to drink 400 grams of nutritive beverage consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a non-nutritive beverage and act as a control for the learned effects.
  Interventions: Behavioral: Learned: Nutritive beverage to Nutritive beverage
- Learned: Non-Nutritive solid to Non-Nutritive solid (Experimental): 15 participants will be randomly assigned to eat 250 grams of non-nutritive solid consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a non-nutritive solid to determine if cephalic phase response changes with learning.
  Interventions: Behavioral: Not Learned: Non-nutritive solid to Nutritive solid
- Learned: Non-Nutritive beverage to Non-Nutritive beverage (Experimental): 15 participants will be randomly assigned to drink 400 grams of non-nutritive beverage consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a non-nutritive beverage to determine if cephalic phase response changes with learning.
  Interventions: Behavioral: Not Learned: Nutritive beverage to Non-nutritive beverage
- Learned: Nutritive solid to Nutritive solid (Experimental): 15 participants will be randomly assigned to eat 250 grams of nutritive solid consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a nutritive solid to determine if cephalic phase response changes with learning.
  Interventions: Behavioral: Not Learned: Non-Nutritive solid to Non-nutritive solid
- Learned: Nutritive beverage to Nutritive beverage (Experimental): 15 participants will be randomly assigned to drink 400 grams of nutritive beverage consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a nutritive beverage to determine if cephalic phase response changes with learning.
  Interventions: Behavioral: Not Learned: Non-nutritive beverage to Nutritive beverage
- Not Learned: Non-Nutritive solid to Non-Nutritive solid (Experimental): 15 participants will be randomly assigned to eat 250 grams of non-nutritive solid consecutively for 2 weeks. After this conditioning, the cephalic phase response of half of these participants will be tested against a non-nutritive solid to determine if cephalic phase response changes with learning.
  Interventions: Behavioral: Not Learned: Non-Nutritive solid to Non-Nutritive Solid

INTERVENTIONS:
Behavioral: Learned: Non-nutritive beverage to Non-nutritive beverage — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a beverage product made with non-nutritive sweetener everyday for two weeks.Half of these participants will then be tested against a non-nutritive beverage.
  Other Names: NNB to NNB
  Arms: Not Learned: Non-nutritive bev to Nutritive bev
Behavioral: Learned: Nutritive solid to Nutritive solid — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a solid food product made with nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a nutritive solid.
  Other Names: NS to NS
  Arms: Not Learned: Nutritive solid to Non-Nutritive solid
Behavioral: Learned: Nutritive beverage to Nutritive beverage — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a beverage product made with nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a nutritive beverage.
  Other Names: NB to NB
  Arms: Not Learned: Nutritive beverage to Non-Nutritive beverage
Behavioral: Not Learned: Non-nutritive solid to Nutritive solid — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a solid food product made with non-nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a nutritive solid.
  Other Names: NNS to NS
  Arms: Learned: Non-Nutritive solid to Non-Nutritive solid
Behavioral: Not Learned: Nutritive beverage to Non-nutritive beverage — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a beverage food product made with nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a non-nutritive beverage.
  Other Names: NB to NNB
  Arms: Learned: Non-Nutritive beverage to Non-Nutritive beverage
Behavioral: Not Learned: Non-Nutritive solid to Non-nutritive solid — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a solid food product made with nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a non-nutritive solid.
  Other Names: NS to NNS
  Arms: Learned: Nutritive solid to Nutritive solid
Behavioral: Not Learned: Non-nutritive beverage to Nutritive beverage — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a beverage food product made with non-nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a nutritive beverage.
  Other Names: NNB to NB
  Arms: Learned: Nutritive beverage to Nutritive beverage
Behavioral: Not Learned: Non-Nutritive solid to Non-Nutritive Solid — For the learning phase of the experiment, random allocation will assign about 15 participants to consume a solid food product made with non-nutritive sweetener everyday for two weeks. Half of these participants will then be tested against a non-nutritive solid.
  Other Names: NNS to NNS
  Arms: Not Learned: Non-Nutritive solid to Non-Nutritive solid

SUMMARY:
This study has two main aims: 1) To determine if ingestion of solid or beverage food forms will change appetite hormone responses, and 2) To determine whether "learning" (defined as 2 week daily consumption) about the metabolic consequence of ingesting solid or beverage foods forms varying in energy alters appetite hormone responses.

Beverage consumption has been implicated in the problem of obesity. However, the exact relationship between beverages, lower appetitive response and lower compensatory dietary responses remains unclear. This study aims to address this gap in the research. For aim 1, the null hypothesis is that the energy in beverage and solid forms will not affect appetite hormonal responses differently. The alternative hypothesis is that exposure to the energy-yielding beverage will elicit a lower appetitive hormone response compared to oral exposure to the solid food form. For aim 2, the null hypothesis is that learning will not change appetite hormone responses. The alternative hypothesis is that learning will decrease appetite hormone responses in the non-energy-yielding beverage more than in the energy-yielding beverage.

DETAILED DESCRIPTION:
The main aims will be studied in 3 phases. In phase 1,the unconditioned cephalic phase responses of participants to nutritive and non-nutritive beverage and solid food forms will be determined. In phase 2, participants will consume a randomly allocated solid food or beverage (either nutritive or non-nutritive) consecutively for 2 weeks. In phase 3, (which will occur immediately after the end of Phase 2), participants will be retested for their cephalic phase responses to determine if there is an effect of learning on appetite hormone response.

ELIGIBILITY:
Inclusion Criteria:

* Body fat percentage > 25% for men and > 32% for women. BMI of 24 kg/m2- 37kg/m2
* No purposeful use of foods or beverages that are sweetened with non-nutritive sweetener > 3 times a week
* No purposeful addition of non-nutritive sweetener to foods and beverages >3 times a week
* No Phenylketonuria (PKU)
* Rate palatability of test load and food sample as greater than 5 on a 9 point category scale.
* Be willing to eat at least 100 grams of carbohydrates for three days prior to each test day
* Self-reported consumer of breakfast and lunch
* Be willing to eat macaroni and cheese during breakfast-lunch hours
* Not taking medications known to influence appetite
* Non-smoker >1 year or more
* Habitual activity pattern over the last 3 months and no plan to change this over the course of the study
* Not on any extreme diet (e.g. Atkins Diet)
* Weight stable (≤ 5 kg change over the last 3 months)
* Not a restrained eater (have a dietary restraint score of <9 on the Three Factor Eating Questionnaire-Restraint section)
* Not a disordered eater (Have a score of <20 in the Eating Attitudes Test-26)
* Have not donated blood for at least 3 months prior to participating in the study
* Indicate no plan to donate blood during, and for three months after the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Appetite Hormone Response | week 1, week 2, week 3, week 4, week 7, week 8, week 9, week 10 (once a week over 136 minutes: 0, 14, 16, 18, 20, 22, 24, 26, 28, 30, 76, 106, 136 minutes)
  Determine the appetite hormone responses to oral exposure of nutritive (energy-yielding) or non-nutritive (non-energy-yielding) sweetener in beverage or solid form. Then, determine whether the appetite hormone responses change after a 2-week learning period.
  Appetite hormones to be measured: Cholecystokinin, Glucagon-Like-Peptide-1, Ghrelin, Insulin, Pancreatic Polypeptide

SECONDARY OUTCOMES:
Change in Appetite | week 1, week 2, week 3, week 4, week 7, week 8, week 9, week 10 (once a week, over 180 minutes: 0, 14, 30, 76, 106, 136, 180 minutes)
  Determining changes in appetite ratings with oral exposure to nutritive or non-nutritive sweetener in beverage or solid food form and lastly with a meal.
Plasma Glucose | week 1, week 2, week 3, week 4, week 7, week 8, week 9, week 10 (once a week, over 136 minutes: 0, 14, 16, 18, 20, 22, 24, 26, 28, 30, 76, 106, 136 minutes)
  Determine the differences in plasma glucose concentration after oral exposure to nutritive or non-nutritive sweetener in beverage or solid food forms and whether there are changes after a 2-week learning period.
Amount of meal ingested | week 1, week 2, week 3, week 4, week 7, week 8, week 9, week 10 (once a week, at 137 minutes to 180 minutes)
  Amount of meal ingested will be determined by presenting a pre-weighted meal and water to the participant at 137 minutes. The meal will be provided in excess of an amount that can be consumed. Participants are asked to eat until comfortably full. The amount ingested will be determined by covertly re-weighing the amount remaining.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States